CLINICAL TRIAL: NCT01606579
Title: An Open-Label, Dose-Escalation Phase I/II Study of PRI-724 for Patients With Advanced Myeloid Malignancies
Brief Title: Safety and Efficacy Study of PRI-724 in Subjects With Advanced Myeloid Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prism Pharma Co., Ltd. (Industry)
Collaborators: inVentiv Health Clinical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRI-724-201
Record Dates: First submitted 2012-05-16; First posted 2012-05-25 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-05

CONDITIONS: Acute Myeloid Leukemia; Chronic Myeloid Leukemia
Keywords: Leukemia; acute myeloid leukemia; AML; chronic myeloid leukemia; CML; MDS; myelodysplastic syndrome; myeloproliferative neoplasia; MPN
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Myelodysplastic Syndromes | interventions — ICG 001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part I (Experimental): Single-agent MTD (or maximum dose to be studied) of PRI-724 will be determined in escalating dose cohorts of Acute Group patients. The MTD cohort will be expanded up to 10 patients to further evaluate tolerability.
  Interventions: Drug: PRI-724
- Part II (Experimental): Single-agent MTD (or maximum dose to be studied) of PRI-724 will be determined in escalating dose cohorts of Non-Acute Group patients. Dosing will begin 2 dose levels below the Part I MTD. The MTD cohort will be expanded up to 10 patients to further evaluate tolerability.
  Interventions: Drug: PRI-724
- Part III Arm A (Experimental): Once the MTD is identified for each arm, that cohort will be expanded to a total of 10 patients each.
  Escalating doses of PRI-724, beginning 2 dose levels below the Part I MTD will be administered in combination with low dose ara-C therapy (20 mg SC BID × 10d q 28d) for AML patients ≥ 65 years of age.
  Interventions: Drug: PRI-724
- Part III Arm B (Experimental): Once the MTD is identified for each arm, that cohort will be expanded to a total of 10 patients each.
  Escalating doses of PRI-724, beginning 2 dose levels below the Part I MTD will be administered in combination with dasatinib (140 mg PO daily) to Acute Group patients with CML-AP or BC.
  Interventions: Drug: PRI-724
- Part III Arm C (Experimental): Once the MTD is identified for each arm, that cohort will be expanded to a total of 10 patients each.
  Escalating doses of PRI-724, beginning 1 dose level below the Part II MTD will be administered in combination with dasatinib (100 mg PO daily) to Non-Acute Group patients with CML-CP.
  Interventions: Drug: PRI-724

INTERVENTIONS:
Drug: PRI-724 — PRI-724
  Arms: Part I; Part II
Drug: PRI-724 — PRI-724 in combination with dasatinib
  Arms: Part III Arm B; Part III Arm C
Drug: PRI-724 — PRI-724 in combination with low dose ara-C therapy
  Arms: Part III Arm A

SUMMARY:
PRI-724 is a new investigational drug being studied to treat subjects with cancer who have advanced myeloid malignancies. PRI-724 is thought to work by blocking the Wnt signaling pathway that cancer cells need to grow and spread (metastasize).

DETAILED DESCRIPTION:
PRI-724 is a new investigational drug being studied to treat subjects with cancer who have advanced myeloid malignancies. PRI-724 is thought to work by blocking the Wnt signaling pathway that cancer cells need to grow and spread (metastasize).

Purpose:

* To test the safety of PRI-724 when taken intravenously (through the vein).
* To observe whether PRI-724 can slow or stop the progression of leukemia.
* To find the Maximum Tolerated Dose (highest safe dose) in the first two parts of the study.
* To find the dose of PRI-724 that should be used in the third part of the study and possible future clinical trials that will study effectiveness and additional safety.
* To test the safety of combining PRI-724 with an approved cancer drug called dasatinib in treating chronic myeloid leukemia (CML).
* To evaluate whether the combination of PRI-724 with the approved cancer drug dasatinib slows or stops the progression of chronic myeloid leukemia (CML).
* To test the safety of combining PRI-724 with an approved cancer drug called Cytarabine in treating acute myelogenous leukemia (AML).
* To evaluate whether the combination of PRI-724 with the approved cancer drug Cytarabine slows or stops the progression of acute myelogenous leukemia (AML).
* To measure how much PRI-724 appears and remains in the blood after infusion.
* To measure several signals called biomarkers associated with cancer in the blood to see if PRI-724 affects those signals.

Study Design:

This will be a single center, open-label escalating-dose cohort study with 3 parts: Part I during which the MTD will be determined in acute group patients; Part II during which the MTD will be determined in non-acute group patients; and Part III during which safety and tolerability of escalating doses of PRI-724 will be assessed in combination with dasatinib for CML patients or low dose ara-C therapy for AML patients ≥ 65 years of age.

ELIGIBILITY:
Inclusion Criteria

1. Patients 18 years or older
2. Part I: Patients with one of the following histologically- or cytologically-proven conditions: relapsed/refractory AML, relapsed/refractory MDS, or advanced CML in AP or BP (i.e., Acute Group patients).
3. Part II: Patients with one of the following documented conditions: CML in CP that is Philadelphia chromosome (Ph)-positive (by cytogenetics) or BCR-ABL1-positive by fluorescent in situ hybridization [FISH], or PCR), as well as resistant to at least 2 FDA-approved tyrosine kinase inhibitors (TKIs); or a myeloproliferative neoplasia which includes: PMF and myelofibrosis secondary to polycythemia vera (PV) and essential thrombocythemia (ET) myelofibrosis (MF) (with intermediate-1, intermediate-2 or high risk disease according to the International Working Group [IWG] prognostic scoring system) (i.e., Non-Acute Group patients).
4. Part III:

   * Arm A: Patients with AML who are 65 years of age or older with refractory or relapsed disease, or who have not received prior therapy but are not eligible to receive intensive frontline chemotherapy (i.e., Acute Group patients);
   * Arm B: Patients with CML in AP or BP, either newly diagnosed or failing TKI therapy (i.e., Acute Group patients);
   * Arm C: Patients with CML in CP after failure of 2 FDA-approved TKIs (i.e., Non-Acute group patients)
5. Performance status 0-2 of the Eastern Cooperative Oncology Group (ECOG) scale
6. Patients must have been off all prior therapy for leukemia except hydroxyurea for 1 week prior to entering this study and recovered from the toxic effects of that therapy
7. Adequate organ function as defined by:

   * Serum creatinine ≤ 2.0 mg/dL or calculated creatinine clearance ≥60 mL/min
   * Total bilirubin ≤2 x ULN (≤5 x ULN if considered due to Gilbert's syndrome or hemolysis)
   * Alanine aminotransferase (ALT) ≤3xULN
8. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
9. Women of childbearing potential and men should practice effective methods of contraception. Women of childbearing potential should have a negative urine or serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin within 7 days prior to the start of PRI 724.

Exclusion Criteria

1. Patients receiving any other investigational agents
2. Patients who are pregnant or breast-feeding
3. Known hypersensitivity to any of the components of PRI-724
4. Pretreatment QTcF interval >470 msec (females) or >450 msec (males)
5. Known active hepatitis B, hepatitis C
6. Serious uncontrolled medical disorder or active systemic infection or current unstable or decompensated medical condition, which makes it undesirable or unsafe for the patient to participate in the study including: New York Heart Association (NYHA) Class 3 or 4, myocardial infarction within 3 months, uncontrolled angina within 3 months, history of clinically significant ventricular arrhythmia, diabetes mellitus with ketoacidosis, or chronic obstructive pulmonary disease (COPD) requiring hospitalization in 6 months prior to the start of treatment with PRI-724.
7. Any other condition, including mental illness or substance abuse deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate, and participate in the study
8. Patients on full dose anticoagulants or any dose of warfarin; patients on prophylactic dose of low-molecular weight or unfractionated heparin are allowed.
9. Patients who have demonstrated intolerance to dasatinib 100 mg daily will not be eligible for Part III/Arm B or C of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-07; Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
DLT (Dose Limiting Toxicity) | 1 year
  Observance of 1 DLT in first 3 patients during 3+3 phase will result in the enrollment of an additional 3 patients.
  Observance of 2+ DLTs in 6 patients during 3+3 phase will result in the next lower dose being expanded.
  Observance of DLTs in 33% of patients in 10 patient MTD expansion will result in the next lower dose being expanded.
  MTD will only be established in a dose level where 0/3 pts or 1/6 pts have a DLT observed in first 2 cycles of therapy.
  Two types of DLTs will be observed: non-hematologic and hematologic.

SECONDARY OUTCOMES:
Preliminary Efficacy Endpoints | 1 year
  The preliminary efficacy endpoints will be changes in the response assessment according to International Working Group Response Criteria for Acute Myeloid Leukemia (AML), European LeukemiaNet Response Criteria for Chronic Myeloid Leukemia (CML), International Working Group Response Criteria for Myelodysplastic Syndromes (MDS) and International Working Group (IWG) consensus criteria for treatment response in myelofibrosis with myeloid metaplasia

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - Emory University / Winship Cancer Institute, Atlanta, Georgia
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas